CLINICAL TRIAL: NCT05479877
Title: A Comparative Clinical and Radiographic Study of Collagen Based Pulpotomy Versus Biodentine Pulpotomy in Children With Cariously Exposed Vital Primary Molars: A Randomized Clinical Trial
Brief Title: A Comparative Clinical and Radiographic Study of Collagen Based Pulpotomy Versus Biodentine Pulpotomy in Children With Cariously Exposed Vital Primary Molars
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nihal Alaa Eldin Mohamed Mostafa Bayoumi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19071991
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Carious Exposure of Pulp
Keywords: pulpotomy; biodentine; collagen
MeSH Terms: interventions — tricalcium silicate; Septodont

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Experimental group) collagen based Pulpotomy (Experimental): (sterile medicated collagen particles, Biofil-AB ,Eucare Pharmaceuticals Pvt. Ltd, Chennai, India)
  Interventions: Drug: sterile medicated collagen particles, Biofil-AB ,Eucare Pharmaceuticals Pvt. Ltd, Chennai, India
- (Control group) Biodentine pulpotomy (Active Comparator): Biodentine (Septodont, Saint-Maur-des-Fossés, France)
  Interventions: Drug: Biodentine (Septodont, Saint-Maur-des-Fossés, France)

INTERVENTIONS:
Drug: sterile medicated collagen particles, Biofil-AB ,Eucare Pharmaceuticals Pvt. Ltd, Chennai, India — Collagen based pulpotomy will be applied (sterile medicated collagen particles, Biofil-AB ,Eucare Pharmaceuticals Pvt. Ltd, Chennai, India)according to the manufacturer's instructions and gently placed over the pulp stumps to a thickness of 2 mm
  Arms: (Experimental group) collagen based Pulpotomy
Drug: Biodentine (Septodont, Saint-Maur-des-Fossés, France) — Biodentine (Septodont, Saint-Maur-des-Fossés, France) will be applied according to the manufacturer's instructions and placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet.
  Arms: (Control group) Biodentine pulpotomy

SUMMARY:
Pulpotomy of vital primary molars is indicated when caries removal results in pulp exposure. Treatment approaches consist of devitalization using formocresol, preservation using ferric sulfate and regeneration of the remaining pulp tissue using mineral trioxide aggregate and recently Biodentine have been utilized.

The ideal pulpotomy medicament would be biocompatible and bactericidal, in addition, to promoting the healing of the root pulp and be compatible with the physiological process of root resorption.

Searching for more pulpotomy agents, Collagen, a protein that's present abundantly in humans, is an important component of connective tissues and performs multiple functions including wound healing.

Enamel and dentin contain Collagen as one of the components in their organic ground matrix.

Collagen has been used widely in dentistry in periodontal and implant therapy as scaffold for preventing the migration of epithelial cells and encouraging wound repopulation by cells with high regenerative potential.

The Collagen available for dental implication is already sterilized and also reinforced with antibiotic particles to efficiently aid in regeneration and repair without any contamination. The collagen particles

DETAILED DESCRIPTION:
Pulpotomy is considered the gold standard procedure for treating cariously exposed pulps in asymptomatic primary teeth. Which is based on the healing ability of the radicular pulp tissue following amputation of the infected coronal pulp.

Mineral trioxide aggregate (MTA) has been recommended as the gold standard for vital pulp therapy; however, it has some disadvantages, such as long setting time, poor handling properties, high cost, and the potential for tooth discoloration. Biodentine (Septodont, Saint-Maur-des-Fossés, France), one of the new-generation, bioactive endodontic cements, has been claimed to have improved properties over MTA.

Biodentine presents high biocompatibility with the dental pulp, it has high antibacterial effects and antifungal activity, has a shorter setting time than MTA as a result of the calcium chloride in the liquid component of Biodentine. It also has higher flexural strength, compressive strength and modulus of elasticity than MTA.

Consequently, Biodentine can be used as a pulp dressing as well as a base material.

Quest is on for newer pulpal medicaments that are biocompatible and capable of healing the dental pulp by producing reparative dentin and/or dentinal bridge in response to various stimuli and surgical exposure.

Collagen has a proven rate of success in the field of dentistry as guided tissue regeneration, root conditioning, hemostatic, and wound dressing agent. It has inherent properties like low immune response and toxicity, ability to promote cellular growth and attachment, homeostasis, and added advantage of antibiotic incorporation.

ELIGIBILITY:
Inclusion Criteria:

* • Children:

  1. Aged 4 to 7, in good general health and medically free.
  2. Cooperative patients who will comply to follow ups.
  3. Parents provided with written informed consent. • Teeth:

  <!-- -->

  1. Bilaterally Carious vital primary molars with reversible pulpitis.
  2. Restorable teeth with no more than 1/3 of root resorption.

Exclusion Criteria:

* • Children:

  1. Children with medical, physical, or mental conditions.
  2. Unable to attend follow up visits. • Teeth:

  <!-- -->

  1. Primary molars with any congenital anomalies.
  2. Previously accessed teeth.
  3. At operative procedure, haemorrhage control is unachievable after pulpotomy.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
absence of internal root resorption | 12 months
  radiographic measurement of internal root resorption

SECONDARY OUTCOMES:
absence of pain and swelling | 12 months
  number of participants with pain and swelling

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT05479877/Prot_000.pdf